CLINICAL TRIAL: NCT00301730
Title: Adoptive Immunotherapy With Costimulated Tumor-Derived T Cells After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Cellular Adoptive Immunotherapy in Treating a Patient Who Has Undergone a Donor Stem Cell Transplant for Breast Cancer That Has Spread to the Lung
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000455626; NCI-05-C-9980; NCI-SE-05-03
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2006-04

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: lung metastases; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — aldesleukin; Trastuzumab; Paclitaxel

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic tumor infiltrating lymphocytes
Biological: trastuzumab
Drug: paclitaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapy, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase I trial is studying how well cellular adoptive immunotherapy works in treating a patient who has undergone a donor stem cell transplant for breast cancer that has spread to the lung.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor response in a patient with persistent metastatic breast cancer after prior allogeneic hematopoietic stem cell transplantation (SCT) treated with tumor-derived, ex vivo expanded and costimulated T-lymphocytes.

Secondary

* Evaluate the immune function of tumor-derived T-lymphocytes and the biology of residual tumor cells present after allogeneic hematopoietic SCT.

OUTLINE: This is a pilot study.

The patient undergoes surgical resection of the accessible lesions from which T cells are isolated, costimulated, and expanded ex vivo to produce the tumor-derived T-lymphocytes (TDTL). Beginning at least 2 weeks after surgery, the patient receives TDTL IV every 4 weeks for up to 5 doses in the presence of disease progression (DP) AND in the absence of ≥ grade 2 graft-versus-host disease. The patient is assessed 4 weeks after every dose.

In case of stable disease, partial response, or complete response, the patient is followed without intervention until DP.

In case of DP after dose 1 or 2 of the TDTL, the patient receives dose 2 or 3 of the TDTL. In case of DP after dose 3 of the TDTL, the patient receives low-dose interleukin-2 subcutaneously (SC) daily for 3 days and dose 4 of the TDTL. In case of DP after dose 4 of the TDTL, the patient receives 1 course of chemoimmunotherapy for cytoreduction and immunomodulation comprising paclitaxel IV over 3 hours once and trastuzumab (Herceptin®) IV over 30-90 minutes once weekly for 3 weeks (the patient may receive gemcitabine hydrochloride, vinorelbine ditartrate, docetaxel, or capecitabine in combination with trastuzumab [Herceptin®] as chemoimmunotherapy at the discretion of the principal investigator); interleukin-2 SC daily for 3 days; and dose 5 of the TDTL. In case of DP after dose 5 of the TDTL, the patient may receive cytotoxic chemotherapy and/or FDA-approved biologic therapy and/or immunotherapy with donor lymphocyte infusions from the same donor used for the prior allogeneic stem cell transplantation.

The patient may undergo core biopsy of the left mediastinal nodule in case of tumor regression of the indexing lesion at anytime OR after receiving dose 5 of the TDTL.

After completion of study treatment, the patient is followed periodically for 5 years.

PROJECTED ACCRUAL: One patient will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IIB HER2/neu-expressing breast cancer 6½ years ago
* Received a T-cell-depleted allogeneic stem cell transplantation (SCT) from a 6/6 HLA-matched sibling donor for refractory metastatic breast cancer
* Developed pulmonary metastases during adjuvant chemotherapy following modified radical mastectomy

  * Pulmonary metastases progressed after prior allogeneic SCT
  * Responded in an objective and measurable manner to prior allogeneic lymphocyte infusion, post-transplantation chemotherapy, and trastuzumab (Herceptin®)
* Disease limited to the thoracic cavity
* Operable tumor with at least 1 cm of surgically accessible lesion

  * Preoperative risk assessment indicating ≤ 5% risk of mortality and < 15% risk of significant morbidity for pulmonary metastasectomy
* Enrolled on protocol CC# 00-C-0119
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy > 6 months
* Negative pregnancy test
* Adequate pulmonary reserve
* Prior graft-versus-host disease (GVHD) ≤ grade 1
* No concurrent GVHD
* No active infection nonresponsive to antimicrobial therapy
* No active psychiatric disorder that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior systemic immunosuppressive therapy
* At least 2 weeks since prior cytotoxic therapy and immunotherapy (e.g. trastuzumab [Herceptin®])
* No concurrent immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Bishop, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States